CLINICAL TRIAL: NCT00065546
Title: Human Requirements for the Nutrient Choline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven Zeisel, Professor of Nutrition and Pediatrics, Director, UNC Nutrition Research Institute, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: DK55865; R01DK055865 (NIH)
Record Dates: First submitted 2003-07-28; First posted 2003-07-31 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Postmenopausal Women
MeSH Terms: interventions — Estrogens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Post-menopausal women randomized to receive estrogen replacement therapy.
  Interventions: Other: Estrogen plus choline depletion diet
- 2 (Placebo Comparator): Post-menopausal women randomized to receive a placebo.
  Interventions: Other: Placebo plus choline depletion diet
- 3 (Experimental): Pre-menopausal women with specific genetic variants.
  Interventions: Other: Pre-menopausal women with SNPs given a low choline diet

INTERVENTIONS:
Other: Estrogen plus choline depletion diet — Post-menopausal subjects receive estrogen and are then challenged with a low choline diet to determine if estrogen protects them from induction of choline deficiency.
  Arms: 1
Other: Placebo plus choline depletion diet — Post-menopausal women are randomized to receive a placebo and are then subjected to a low choline diet to determine if clinical signs of choline deficiency can be induced.
  Arms: 2
Other: Pre-menopausal women with SNPs given a low choline diet — Pre-menopausal women with specific genetic polymorphisms in genes related to choline metabolism are placed on a choline depletion diet to determine if the SNPs increase or decrease the risk of diet-induced choline deficiency.
  Arms: 3

SUMMARY:
The purpose of this study is to increase our understanding of how much choline humans need to get from their diet. Choline is an essential nutrient found in many foods, including eggs and milk. In addition to dietary sources, choline can be made in the liver. Choline is important in making membranes or wrappers for all the cells in the body and for making chemicals that allow nerve cells to work properly. In a previous study we found that the dietary requirement for choline varies greatly from person to person. This was caused, in part, by how much estrogen a person has and their genetic makeup. We are conducting this study to explore how estrogen levels and specific differences in genes influence choline requirements so that we can refine the dietary recommendations for this nutrient.

DETAILED DESCRIPTION:
Choline is an essential nutrient essential used for the structural integrity and signaling functions of cell membranes, cholinergic neurotransmission, and lipid transport/metabolism. Choline is obtained from the diet and from endogenous biosynthesis catalyzed by the enzyme phosphatidylethanolamine N-methyltransferase (PEMT). The major premise for this proposal is that humans require a dietary source of choline and that this requirement has significant individual variation and is modulated by estrogen and common genetic polymorphisms. The promoter of the PEMT gene is estrogen responsive, and we hypothesize that estrogen status influences the dietary requirement for choline. We identified other common single nucleotide polymorphisms (SNPs) that increase or decrease the likelihood that a human will develop organ dysfunction when fed a low choline diet. Experiments are proposed that will refine our understanding of estrogen-mediated induction of the PEMT promoter; determine whether postmenopausal women treated with estrogen have a decreased susceptibility to developing organ dysfunction associated with choline deficiency; determine the prevalence of SNPs that increase susceptibility to choline deficiency in the population and examine dietary choline requirements in humans with these SNPs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoker
* BMI between 18 and 34
* Normal mammogram in last 12 months (post-menopausal women only)

Exclusion Criteria:

* Hormone or estrogen therapy
* Allergic to soy, eggs, wheat
* History of breast, uterine, or other estrogen-dependent cancer
* Liver or kidney problems
* History of circulation, bleeding, or blood-clotting disorder
* Anemia or evidence of iron overload
* Hyperthyroidism, neurological disorder, or autoimmune disease
* Diabetes controlled by insulin
* Positive serology for HIV or Hepatitis B or C
* Alcohol or illegal drug misuse/abuse
* Pacemaker, aneurysm clip, cardiac heart valve, mechanical devices/implants
* Other metal in body (i.e. injured by a BB, shrapnel, or metallic object)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Evidence of liver or muscle dysfunction (based on elevations in CPK, AST, ALT), or increased liver fat (measured by liver MRI) | Labs measured every 3-4 days throughout 62-day trial. Liver MRI performed on study days 1, 10, 31, 52, 62.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Zeisel, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Leslie M Fischer, PhD, MPH, RD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] da Costa KA, Corbin KD, Niculescu MD, Galanko JA, Zeisel SH. Identification of new genetic polymorphisms that alter the dietary requirement for choline and vary in their distribution across ethnic and racial groups. FASEB J. 2014 Jul;28(7):2970-8. doi: 10.1096/fj.14-249557. Epub 2014 Mar 26. PMID 24671709
- [Derived] da Costa KA, Sanders LM, Fischer LM, Zeisel SH. Docosahexaenoic acid in plasma phosphatidylcholine may be a potential marker for in vivo phosphatidylethanolamine N-methyltransferase activity in humans. Am J Clin Nutr. 2011 May;93(5):968-74. doi: 10.3945/ajcn.110.011064. Epub 2011 Mar 16. PMID 21411618
- [Derived] Fischer LM, da Costa KA, Kwock L, Galanko J, Zeisel SH. Dietary choline requirements of women: effects of estrogen and genetic variation. Am J Clin Nutr. 2010 Nov;92(5):1113-9. doi: 10.3945/ajcn.2010.30064. Epub 2010 Sep 22. PMID 20861172